CLINICAL TRIAL: NCT05260814
Title: Comparison of Two Oral Hygiene Routines on the Glycemic Control for Type 2 Diabetes Patients With Chronic Periodontitis. A Prospective Randomized Controlled Clinical Trial
Brief Title: Comparison of Two Oral Hygiene Routines on the Glycemic Control for Type 2 Diabetes Patients With Chronic Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Harvard School of Dental Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB21-0148
Record Dates: First submitted 2022-01-25; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Periodontal Diseases; Diabetes Mellitus
Keywords: periodontitis; diabetes mellitus; electric toothbrush
MeSH Terms: conditions — Periodontal Diseases; Diabetes Mellitus; Periodontitis

STUDY DESIGN:
Intervention Model Description: Randomized control clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Scaling and root planing and oral hygiene instructions with use of manual tools
- Experimental (Experimental): Scaling and root planing, oral hygiene instructions with use of Sonicare Diamond Clean Smart®.
  Interventions: Device: Electric toothbrush with smart phone app

INTERVENTIONS:
Device: Electric toothbrush with smart phone app — Scaling and root planing, oral hygiene instructions with use of Sonicare Diamond Clean Smart®.
  Arms: Experimental

SUMMARY:
This study aims to compare two common oral hygiene routines on the improvement of glycemic control and oral health parameters in moderate to severe periodontitis patients with uncontrolled type 2 diabetes (T2DM).

It is currently unclear if one oral hygiene routine is more effective than the other. The two routines being compared are:

Group 1: Scaling and root planing + oral hygiene routine with use of an electric toothbrush (Sonicare Diamond Clean Smart ®) along with its mobile app Group 2: Scaling and root planing + oral hygiene routine with use of manual toothbrush

The specific aims of the study are:

Aim 1: To assess the impact of Sonicare Diamond Clean Smart ® use on the glycemic control as an adjunct to scaling and root planing and oral hygiene instructions for T2DM patients with moderate to severe periodontitis patients.

Aim 2: To assess oral health parameters which include clinical measurements and immune-inflammatory cytokines.

DETAILED DESCRIPTION:
Background Periodontitis is among the most prevalent chronic diseases in the world and it affects more than 50% of Americans. On the other hand, type 2 diabetes mellitus (T2DM) is a major public health concern, affecting 347 million adults worldwide. This number will likely double by the year 2030 with diabetes-related health care expenditure amount to 15%. The relationship between periodontal diseases and diabetes has been well-established. Treatment of periodontal diseases improves diabetes outcomes.

To treat and prevent gingivitis as well as periodontal disease, microbial plaque biofilm control is essential. A classic study done in 1965 clearly demonstrated the relationship between plaque accumulation when subjects stopped brushing and the development of gingivitis in humans. Adherence to oral hygiene care by the patient is an important part in the maintenance of periodontal health. Oral hygiene reinforcement through repeated oral hygiene instructions as well as psychological interventions have shown to have positive effects on oral hygiene improvement.

Rapid communication, health information access and monitoring have been made possible through the various innovations in mobile device. However, at present, no studies have investigated the impact of the incorporation of electric-toothbrush and smart device for self-monitoring for the periodontal treatment outcomes on diabetes patients. It is currently unclear whether a toothbrush with smartphone application that incorporates self-efficacy and behavioral modification will result in improved clinical parameters, reduction in inflammation and periodontal pathogens in blood as well as glycemic control for these patients.

Specific Aims This study aims to investigate the efficacy of Sonicare Diamond Clean Smart ® on the improvement of glycemic control and oral health parameters in moderate to severe periodontitis patients with uncontrolled type 2 diabetes (T2DM).

The primary objective of this study is to assess the efficacy of Sonicare Diamond Clean Smart ® on the glycemic control as an adjunct to scaling and root planing and oral hygiene instructions for T2DM patients with moderate to severe periodontitis patients.

The secondary objective is to assess oral health parameters which include clinical measurements and immune-inflammatory cytokines.

The two groups being compared are:

• Experiment group: Scaling and root planing, oral hygiene instructions with use of Sonicare Diamond Clean Smart®.

• Control group: Scaling and root planing and oral hygiene instructions with use of manual tools.

Study Design The study protocol will be submitted for approval by the Harvard Medical School IRB committee. The study will begin following IRB approval. Forty subjects (40) with moderate to severe periodontal disease and diagnosed with uncontrolled type 2 diabetes mellitus (T2DM) will be recruited into study. Of these, twenty will be randomized into experimental group while the other twenty will be randomized into control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 35 or above.
* A minimum of 16 teeth (not including third molars) exists.
* Diagnosis of moderate to severe periodontitis (stage-II to stage-III chronic periodontitis)
* Clinical attachment loss ≥2mm and probing depths of ≥ 5mm in two or more quadrants in the mouth.
* A minimum of 50% of sites exhibiting bleeding on probing.
* FMX shows bone loss at least 15% ~50% at least one site.
* Diagnosis of type 2 diabetes mellitus (T2DM) with last HbA1c level > 7%
* Willing to participate in the study and follow all visits.
* Have mobile phones compatible with use of the Philips Sonicare Digital App

Exclusion Criteria:

* Systemic condition requiring antibiotic prophylaxis prior to any invasive procedure
* Systemic disease other than diabetes that would impair healing such as patients on immunosuppression meds, with autoimmune disease, chemo/radiation therapy within the last 10 years
* Subjects with dental implants
* Subjects with implanted pacemakers/defibrillators
* Subjects on prescription for blood thinners
* Antibiotic use within the last 8 weeks (if subjects get placed on antibiotics due to infection for other unrelated health issues during the study period, this will be recorded)
* Long-term use of non-steroidal anti-inflammatory drugs (NSAIDs)
* Pregnant/nursing
* Smokers
* Fully edentulous in either Maxilla or Mandibular
* Previous periodontal treatment in the last 6 months
* Do not have mobile phones for use with the digital app from Philips

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
changes in HbA1c | 12 months
  To assess the impact of Sonicare Diamond Clean Smart ® use on the glycemic control as an adjunct to scaling and root planing and oral hygiene instructions for T2DM patients with moderate to severe periodontitis patients.

SECONDARY OUTCOMES:
probing pocket depth changes | 12 months
  To assess oral health parameters which include clinical measurements and immune-inflammatory cytokines.
cytokine changes | 12 months
  To assess oral health parameters which include clinical measurements and immune-inflammatory cytokines.

IPD SHARING:
Plan to Share IPD: Undecided